CLINICAL TRIAL: NCT02587078
Title: Volume Therapy With Crystalloids and Colloids
Brief Title: Volume Therapy With Crystalloids and Colloids and Hemodynamic Monitoring in Patients With Severe Sepsis
Acronym: VOMOSEP
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: treatment substance not labled for sepsis anymore
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-VS01-01; 2012-000331-30 (EudraCT Number)
Record Dates: First submitted 2014-12-10; First posted 2015-10-27 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-03

CONDITIONS: Severe Sepsis
Keywords: Haemodynamic stabilization
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Volulyte (Active Comparator): Patients who meet the inclusion criteria (at Screening, see below for definition) will be randomized immediately in a ratio of 1:1 to either intravenous Volulyte® or Jonosteril® for fluid resuscitation (on RAND). Fluid resuscitation with study drug will be started immediately in order to reach initial hemodynamic stabilization.
  Interventions: Drug: Jonosteril
- Jonosteril (Active Comparator): Patients who meet the inclusion criteria (at Screening, see below for definition) will be randomized immediately in a ratio of 1:1 to either intravenous Volulyte® or Jonosteril® for fluid resuscitation (on RAND). Fluid resuscitation with study drug will be started immediately in order to reach initial hemodynamic stabilization.
  Interventions: Drug: Volulyte

INTERVENTIONS:
Drug: Volulyte — Patients who meet the inclusion criteria (at Screening, see below for definition) will be randomized immediately in a ratio of 1:1 to either intravenous Volulyte® or Jonosteril® for fluid resuscitation (on RAND). Fluid resuscitation with study drug will be started immediately in order to reach initial hemodynamic stabilization.
  Arms: Jonosteril
Drug: Jonosteril — Patients who meet the inclusion criteria (at Screening, see below for definition) will be randomized immediately in a ratio of 1:1 to either intravenous Volulyte® or Jonosteril® for fluid resuscitation (on RAND). Fluid resuscitation with study drug will be started immediately in order to reach initial hemodynamic stabilization.
  Arms: Volulyte

SUMMARY:
The primary alternative hypothesis is that less time (minutes) is required, to achieve the initial hemodynamic stabilization, with Volulyte® compared to Jonosteril®.

* H01: Minutes with Volulyte® ≥ Minutes with Jonosteril®
* H11: Minutes with Volulyte® < Minutes with Jonosteril®

DETAILED DESCRIPTION:
Comparative, multicenter, active-controlled, parallel-group, double-blind, randomized study.

Patients who meet the inclusion criteria (at Screening, see below for definition) will be randomized immediately in a ratio of 1:1 to either receive intravenous Volulyte® or Jonosteril® for fluid resuscitation (on RAND). Fluid resuscitation with study drug will be started immediately in order to reach initial hemodynamic stabilization. Assessment of the effects of fluid resuscitation to achieve the primary and secondary endpoints will be performed up to 24 hours following the randomization.

Initial hemodynamic stabilization is defined as normalization of mean arterial pressure (MAP), central venous oxygen saturation (ScvO2) and PPV (pulse pressure variation) or response to PLR (passive leg rising) as defined below and maintaining this normalization over a period of 1 hour, with no increase in the infusion of vasopressors, or inotropic therapy and with ≤ 250ml of additional study drug administration within this 1 hour. The normalization of the parameters MAP and PPV (pulse pressure variation) or PLR (passive leg rising) and ScvO2 is defined as follows:

* MAP: ≥ 65 mmHg
* ScvO2: ≥ 70%
* PPV: ≤ 12% (premise: sinus rhythm, no spontaneous breathing efforts and mechanical ventilation with VT: 5 - < 6 ml/kg).

If PPV is not applicable, response to PLR-manoeuvre is used (see below).

● PLR: < 10% change in cardiac output (CO)

ELIGIBILITY:
Inclusion Criteria:

1. Prior written informed consent of the patient. If this is not possible, it will be necessary for the investigator to obtain initial informed consent according to the requirements. The legally authorized representative has to provide the written informed consent or in his absence a declaration for inclusion in an emergency situation is to be signed by a consultant physician who is not involved in the study and who is independent of the investigational team. If the patient dies following the inclusion in the clinical trial based on the consulting physician´s vote and no legally authorized representative is available / able to give informed consent, no additional informed consent will be needed and the consultant physician´s vote will be considered sufficient.
2. Male or female patient aged 18 years or older
3. Presence of severe sepsis defined as:

   * Sepsis due to a known or suspected infection with two or more of the modified systemic inflammatory response syndrome (SIRS) criteria (46).

     * Temperature (> 38°C or < 36°C)
     * Heart rate (> 90 beats / minute)
     * Respiratory rate (>20 breaths / minute) or arterial carbon dioxide (PaCO2) < 32 mmHg (< 4.3 kPa)
     * White blood cells (WBC) > 12.000 cells/mm3, < 4000 cells/mm3, or > 10% immature (band) forms
   * Severe sepsis for less than 24 hours with at least one of the following characteristics:

     * Ratio of partial pressure of oxygen to the fraction of inspired oxygen (PaO2/FiO2) < 250
     * Arterial pH < 7.3 or serum lactate level > 1.5 × ULN (upper limit of normal)
     * Hypotension: Inadequately fluid resuscitated patients with a systolic blood pressure ≤ 90 mmHg or MAP ≤ 70 mmHg, or adequately fluid resuscitated patients requiring vasopressors to maintain blood pressure within normal ranges
     * Urine output < 0.5 ml/kg/hour (patients who are inadequately fluid resuscitated)
     * Platelet count < 80.000/ mm3
     * Acute alteration of mental status
4. Requirement for fluid resuscitation as defined by the measured hemodynamic parameters MAP, ScvO2 and PPV or PLR.

Exclusion Criteria:

1. Volume expansion with a dosage of HES administered prior to randomization rendering a patient unsuitable for inclusion based on the treating physician´s discretion in consideration of the suggested maximal dose/day.
2. Known volume expansion with any dosage of HES 200.000 prior to inclusion during the actual hospital admission.
3. Participation in another clinical study with an investigational drug or an investigational medical device within 30 days before screening or planned during the study period.
4. Known hypersensitivity to any components of the investigated solutions.
5. Known pregnancy; female patients must be surgically sterile; or postmenopausal for at least two years; or if of childbearing potential must have a negative serum or urine dipstick pregnancy test (if a test result is not available at the time of randomization, a patient may be randomized and treated initially, however, has to be withdrawn immediately from the study as soon as the test result becomes available and is positive).
6. Known serum creatinine > 300 μmol/L, corresponding to 3.4 mg/dL (if a serum creatinine value is not available at the time of randomization or an available value is older than 24 hours, a patient may be randomized and treated. If a creatinine value of > 300 μmol/L becomes available later, treatment with the study drug may be continued if the risk/benefit ratio for the individual patient is regarded as positive by the investigator.)
7. Known history of chronic renal failure (hemodialysis)
8. Anuria lasting more than 8 hours (<50ml urine output / 8 hours) despite fluid resuscitation prior to randomization.
9. Requirement for renal support (either continuous or discontinuous techniques, including intermittent hemodialysis, hemofiltration and hemodiafiltration)
10. History of known hemostatic disorders with clinical bleeding (hemophilia and known or suspected Willebrand disease)
11. Burns >20% of body surface
12. State of brain death
13. Known co-morbidities: Hematologic malignant disorders, neutropenia (polymorphonuclear leukocytes [PMN] < 500/mm3), proven liver cirrhosis, Aquired immunodeficiency syndrome (AIDS) Expected requirement for concomitant cancer therapy (e.g. chemotherapradiotherapy or surgery) from randomization until Day 4 Requirement for concomitant cancer therapy (e.g. chemotherapy, radiotherapy or surgery) from randomization until Day 4
14. Known fluid overload (EVLWI > 10 ml/kg BW)
15. Need for fluid restriction
16. Refractory septic shock defined as severe sepsis with hypotension unresponsive to adequate fluid resuscitation, along with the presence of hypoperfusion abnormalities or organ dysfunction as defined by Bone et al., 1992. Patients receiving inotropic or vasopressor agents may no longer be hypotensive by the time they manifest hypoperfusion abnormalities or organ dysfunction, yet they would still be considered to have septic shock. Patients treated with low dose vasopressors are not excluded provided they are responsive to fluid resuscitation as demonstrated by an individual fluid challenge. Patients receiving norepinephrine (noradrenaline) or epinephrine (adrenaline) at a dose > 0.5 μg/kg/min or dopamine at a dose > 15 μg/kg/min at the timepoint of Screening are not eligible for the study.
17. Intracranial bleeding
18. Any condition rendering a patient unsuitable for inclusion based on the treating physician´s discretion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is defined as the fraction of patients who achieved initial hemodynamic stabilization during the first 6 hours after randomisation. | During the first 6 hours

SECONDARY OUTCOMES:
Time needed for achievement of initial hemodynamic stabilization during the first 24 hours after randomization. | during the first 24 hours after randomization.

IPD SHARING:
Plan to Share IPD: Undecided